CLINICAL TRIAL: NCT00093379
Title: A Phase II Study of Capecitabine (Xeloda)/Oxaliplatin (Eloxatin) With Concomitant Radiotherapy (XRT), XELOX/RT in Squamous Cell Carcinoma of the Anal Canal
Brief Title: Capecitabine, Oxaliplatin, and Radiation Therapy in Treating Patients With Stage II or Stage III Anal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0874; P30CA016672 (NIH); MDA-2003-0874 (Other: UT MD Anderson Cancer Center); SANOFI-MDA-2003-0874; CDR0000380771 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Anal Cancer
Keywords: stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; squamous cell carcinoma of the anus; Capecitabine; Xeloda; Oxaliplatin; Eloxatin; Radiotherapy; XRT
MeSH Terms: conditions — Anus Neoplasms | interventions — Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine + Oxaliplatin + XRT (Experimental): Capecitabine (825 mg/m^2 twice a day, Monday-Friday during weeks 1, 2, 4, and 5) and Oxaliplatin (50 mg/m^2, Days 1, 8, 22, 29) during the duration of radiation therapy only. Radiotherapy once daily on days 1-3, 6-10, 13-17, 20-24, 27-31, 34-38, and 41-42. Participants with T3-4 lesions undergo radiotherapy once daily on days 43 and 44. The final dose of radiation therapy determined by the T stage of the primary tumor. Radiotherapy = XRT.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiation Therapy (XRT)

INTERVENTIONS:
Drug: Capecitabine — 825 mg/m^2 orally twice a day (BID), Mon-Fri during weeks 1, 2, 4, and 5.
  Other Names: Xeloda
Drug: Oxaliplatin — 50 mg/m^2 by vein (IV) over 2 hours on days 1, 8, 22, and 29.
  Other Names: Eloxatin
Radiation: Radiation Therapy (XRT) — Undergo radiotherapy* once daily on days 1-3, 6-10, 13-17, 20-24, 27-31, 34-38, and 41-42. *Patients with T3-4 lesions undergo radiotherapy once daily on days 43 and 44.
  Other Names: XRT; RT; Radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Capecitabine may stop the growth of tumor cells by stopping blood flow to the tumor. Radiation therapy uses high-energy x-rays to damage tumor cells. Capecitabine and oxaliplatin may make tumor cells more sensitive to radiation therapy. Combining capecitabine and oxaliplatin with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine and oxaliplatin together with radiation therapy works in treating patients with stage II or stage III anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine time to treatment failure in patients with stage II-IIIB squamous cell carcinoma of the anal canal treated with capecitabine, oxaliplatin, and radiotherapy (i.e. Capecitabine (Xeloda)/Oxaliplatin (Eloxatin) With Concomitant Radiotherapy (XRT) shortened to XELOX/XRT).
* Determine the toxic effects of this regimen in these patients.

Secondary

* Determine the complete response rate in patients treated with this regimen.
* Determine 2-year local regional control in patients treated with this regimen.
* Determine 2-year colostomy-free survival in patients treated with this regimen.
* Determine 2-year median overall survival in patients treated with this regimen.
* Determine 2-year progression-free survival in patients treated with this regimen.

OUTLINE: Patients receive oral capecitabine* twice daily on days 1-2, 6-10, 20-24, 27-31, and 41-42, and undergo radiotherapy* once daily on days 1-3, 6-10, 13-17, 20-24, 27-31, 34-38, and 41-42. Patients also receive oxaliplatin intravenous (IV) over 2 hours on days 1, 8, 22, and 29. Treatment continues in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients with T3-4 lesions also receive oral capecitabine twice daily and undergo radiotherapy once daily on days 43 and 44.

Patients are followed at 4-6 and 12 weeks and then periodically thereafter.

PROJECTED ACCRUAL: A total of 71 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated patients with histologically proven squamous cell carcinoma of the anal canal.
2. American Joint Committee on Cancer (AJCC) stage II-IIIB (TX 1-4, NX, MO).
3. Age >/= 16 yrs old.
4. Eastern Cooperative Oncology Group (ECOG) Performance Scale (PS) 0-1.
5. Adequate organ function including: Absolute neutrophil Count (ANC) >/= 1,500/uL, Platelets >/= 100,000/uL, Total bilirubin </= 1.5 * upper limit of normal (ULN), aspartate aminotransferase (AST or SGOT)/alanine aminotransferase (ALT or SGPT) </= 3 * ULN, Creatinine </= 1.5mg/dL or Creatinine Clearance (CrCL) >/= 50 cc/min.
6. Patients may have measurable or non-measurable disease. Patients with measurable disease, as defined by the modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria, have at least one lesion that can be accurately measured in at least one dimension with longest diameter to be recorded >/= 20 mm using conventional techniques or >/= 10 mm with spiral CT scan (with minimum lesion size no less than double the slice thickness). Lesions seen on colonoscopy or barium studies are not considered measurable lesions.
7. A negative pregnancy test in all women of child-bearing potential, within two weeks of initiating treatment.
8. The effects of oxaliplatin and capecitabine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because cytotoxic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
9. Ability to understand and the willingness to sign the written informed consent/authorization document.

Exclusion Criteria:

1. Prior chemotherapy with oxaliplatin, capecitabine, or 5-fluorouracil.
2. Prior radiation to the pelvis.
3. Prior surgery for anal cancer excluding prior biopsy.
4. Known history of dihydropyrimidine (DPD) deficiency.
5. Known history of hypersensitivity to platinum-containing compounds.
6. Peripheral neuropathy of >/= grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) 3.0.
7. Calculated creatinine clearance (CrCl) < 50 cc/min.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit adherence with study requirements.
9. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation.
10. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with oxaliplatin or capecitabine, breast feeding should be discontinued.
11. Because of the known interaction of capecitabine and coumadin, patients taking coumadin will be ineligible. Patients will be requested to discontinue coumadin and utilize Lovenox if agreeable. Patients must have discontinued coumadin for 7 days before initiating therapy.
12. No prior malignancies (excluding non-melanomatous skin neoplasms) over the past 5 years.
13. HIV-positive patients receiving combination anti-retroviral therapy are excluded from this study because of possible pharmacokinetic interactions with capecitabine or oxaliplatin. This exclusion is for patient safety since patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, and because very few HIV-positive anal canal cancer patients are seen at this institution. This hinders us from accruing enough patients to adequately test the safety of this regimen in this population.
14. Patients with symptomatic pulmonary fibrosis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Eng, MD, Study Chair — M.D. Anderson Cancer Center; Christopher H. Crane, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- [Derived] Eng C, Jacome AA, Das P, Chang GJ, Rodriguez-Bigas M, Skibber JM, Wolff RA, Qiao W, Xing Y, Sethi S, Ohinata A, Crane CH. A Phase II Study of Capecitabine/Oxaliplatin With Concurrent Radiotherapy in Locally Advanced Squamous Cell Carcinoma of the Anal Canal. Clin Colorectal Cancer. 2019 Dec;18(4):301-306. doi: 10.1016/j.clcc.2019.06.003. Epub 2019 Jul 2. PMID 31350201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period: April 16, 2004 to May 12, 2009. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Capecitabine + Oxaliplatin + XRT: Capecitabine (825 mg/m^2 twice a day, Monday-Friday during weeks 1, 2, 4, and 5) and Oxaliplatin (50 mg/m^2, Days 1, 8, 22, 29) during the duration of radiation therapy only. Radiotherapy (XRT) once daily on days 1-3, 6-10, 13-17, 20-24, 27-31, 34-38, and 41-42. Participants with T3-4 lesions undergo radiotherapy once daily on days 43 and 44. The final dose of radiation therapy determined by the T stage of the primary tumor.
Period: Overall Study
Arm/Group | Capecitabine + Oxaliplatin + XRT
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine + Oxaliplatin + XRT
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 55 [39 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Failure Free Survival
Description: Treatment failure defined as: Biopsy proven residual disease identified 12 -14 weeks after the conclusion of chemoradiation therapy, Treatment-related mortality or Disease recurrence.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Capecitabine + Oxaliplatin + XRT
Number analyzed (Participants) | 20
participants | 20

2. Secondary Outcome: Number of Participants With Complete Response at 2 Years
Description: Response determined by computed tomography (CT)/magnetic resonance imaging (MRI), digital rectal examination, and proctoscopy, and a biopsy performed for clinical suspicion of residual or progressive disease. Response Evaluation Criteria in Solid Tumors (RECIST) where evaluation of target lesions Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 2 Years
Population: Three (3) participants were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Capecitabine + Oxaliplatin + XRT
Number analyzed (Participants) | 17
participants | 16

3. Secondary Outcome: Number of Participants With 2-year Colostomy-Free Survival
Description: Colostomy-free survival reported as number of participants who did not develop local recurrence or require salvage resection with colostomy.
Time Frame: 2 Years with median study follow up of 19 months
Measure: Number; unit: participants
Arm/Group | Capecitabine + Oxaliplatin + XRT
Number analyzed (Participants) | 20
participants | 20

4. Secondary Outcome: 2-year Local Regional Control
Time Frame: 2 Years
Reporting Status: Not Posted

5. Secondary Outcome: 2-Year Median Overall Survival
Time Frame: 2 Years
Reporting Status: Not Posted

6. Secondary Outcome: Number of Participants With Progression-Free Survival at 2-Year
Time Frame: 2 Years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years and 9 months
Arm/Group | Capecitabine + Oxaliplatin + XRT
Serious Adverse Events (participants affected / at risk) | 20/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Oxaliplatin + XRT (N=20)
•Increased Aspartate aminotransferase (AST, SGOT) (Blood and lymphatic system disorders) | 1
Dehydration (General disorders) | 1
Allergic Reaction Including Drug Fever (Infections and infestations) | 1
Dermatitis (Chemoradiation) (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Radiation) (Skin and subcutaneous tissue disorders) | 4
Diarrhea (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain (General disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Oxaliplatin + XRT (N=20)
Allergic Reaction Including Drug Fever (Metabolism and nutrition disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Increased Alanine aminotransferase (ALT, SGPT) (Blood and lymphatic system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 6
Increased Aspartate aminotransferase (AST, SGOT) (Blood and lymphatic system disorders) | 3
Elevated Bilirubin (Blood and lymphatic system disorders) | 1
Bloody Stool (Gastrointestinal disorders) | 1
Blurred Vision (Eye disorders) | 1
Bowel Movement, Changes (Gastrointestinal disorders) | 1
Blood urea nitrogen (BUN) Increase (Renal and urinary disorders) | 1
Burn (Injury, poisoning and procedural complications) | 1
Cold Intolerance (Nervous system disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Cystitis (Reproductive system and breast disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Dermatitis (Chemoradiation) (Skin and subcutaneous tissue disorders) | 8
Dermatitis (Radiation) (Skin and subcutaneous tissue disorders) | 4
Dermatology/Skin (Other) (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Fatigue (General disorders) | 9
Fever Without Neutropenia (Infections and infestations) | 5
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal (Other) (Gastrointestinal disorders) | 3
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 1
Elevated Hemoglobin (Blood and lymphatic system disorders) | 3
GI Hemorrhage (Gastrointestinal disorders) | 4 — Hemorrhage, GI (Anus): 1 participant Hemorrhage, GI (Rectum): 3 participants
Hot Flashes (Reproductive system and breast disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Blood and lymphatic system disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Infection (Other) (Infections and infestations) | 2
Infection Clinical with Grade 3-4 ANC (Infections and infestations) | 2 — Infection with Grade 3-4 Absolute Neutrophil Count (ANC); Urinary Tract, Vagina
Infection with Normal ANC (Infections and infestations) | 3 — Urinary Tract, Vagina, Vulva
Insomnia (Psychiatric disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Metabolic Problem (Metabolism and nutrition disorders) | 1
Mucositis (Gastrointestinal disorders) | 3
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Issue (Other) (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Neurological Issues (Other) (Nervous system disorders) | 3
Neuropathy: Cranial (Nervous system disorders) | 1 — Cn X Motor-Palate, Pharynx, Larynx
Increased Neutrophils (Absolute neutrophil count (ANC)/Absolute Granulocyte Count (AGC) (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 20 — Abdomen, Anus, Chest Wall, Eye, Head/Headache, Muscle, Neck, Perineum, Rectum, Tumor, Urethra, Rectal and other areas.
Proctitis (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Dermatitis (Radiation) (Skin and subcutaneous tissue disorders) | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1
Rectal Bleeding (Gastrointestinal disorders) | 2
Renal/Genitourinary (Other) (Renal and urinary disorders) | 5
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Rigors/Chills (General disorders) | 1
Sinus Tachycardia (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Gastrointestinal disorders) | 1
Stricture/Stenosis, GI (Rectum) (Gastrointestinal disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 2
Telangiectasia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Ulcer, GI (Rectum) (Gastrointestinal disorders) | 1
Vaginal Bleeding (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Vaginal Dryness (Reproductive system and breast disorders) | 2
Vaginal Stenosis (Reproductive system and breast disorders) | 1
Vaginitis (Reproductive system and breast disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Watery Eye (Eye disorders) | 1
Weight Loss (Gastrointestinal disorders) | 6
Yeast Infection (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No